CLINICAL TRIAL: NCT01924481
Title: Effects of a Cocoa Shot on the Human Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00023752
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Caffeine; Flavonoids
Keywords: Caffeine; Flavonoids; MRI; Brain blood flow; Cognition; Perfusion; Resting functional magnetic resonance imaging (fMRI)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low theobromine & low caffeine (Experimental): Drink 1
  Interventions: Dietary Supplement: Low caffeine; Dietary Supplement: low theobromine
- low theobromine & high caffeine (Experimental): Drink 2
  Interventions: Dietary Supplement: High Caffeine; Dietary Supplement: low theobromine
- high theobromine & low caffeine (Experimental): Drink 3
  Interventions: Dietary Supplement: Low caffeine; Dietary Supplement: High theobromine
- no theobromine & high caffeine (Active Comparator): Drink 4
  Interventions: Dietary Supplement: High Caffeine; Dietary Supplement: No theobromine

INTERVENTIONS:
Dietary Supplement: High Caffeine
  Arms: low theobromine & high caffeine; no theobromine & high caffeine
Dietary Supplement: Low caffeine
  Arms: high theobromine & low caffeine; low theobromine & low caffeine
Dietary Supplement: High theobromine
  Arms: high theobromine & low caffeine
Dietary Supplement: low theobromine
  Arms: low theobromine & high caffeine; low theobromine & low caffeine
Dietary Supplement: No theobromine
  Arms: no theobromine & high caffeine

SUMMARY:
The Hershey Company is interested in investigating the effects of various chocolate beverages on brain physiology and cognitive function. The main substances in the drinks that are known to influence the brain are caffeine (and related chemicals such as theobromine) and flavonoids. Flavonoids are chemical found in plants and are most commonly associated with antioxidant activity. Caffeine, chemicals related to caffeine, and flavonoids are all naturally occurring and all potentially alter brain physiology. This study will evaluate changes in brain blood flow and cognition following the consumption of drinks with various combinations of the Primary Ingredients. Caffeine is likely to have peak effects within 1-hour of ingesting the chocolate while the flavonoids are likely to have peak effects 3-4 hours after ingestion. The study proposed here will evaluate ingredients in a 4-arm cross-over double-blind design in an attempt to understand the differential effects of these compounds in chocolate drinks.

ELIGIBILITY:
Inclusion Criteria:

* Consume 200-600 mg caffeine daily
* Willing and capable of signing the informed consent
* Willing to attend 4 testing sessions that will take 4-6 hours each AND will be at least 7 days apart
* Willing to abstain from caffeine for 24 hours before each testing session
* Willing to and able to have MRIs

Exclusion Criteria:

* As determined from the medical screening session

  * active neurological dysfunction (such as a major Axis I psychopathology, Alzheimer's disease, Parkinson's disease, prior history of stroke, epilepsy, or serious central nervous system (CNS) trauma)
  * attention deficit hyperactivity disorder (ADHD)
  * migraines
  * hypertension
  * diabetes
  * peripheral vascular disease
  * taking vasoactive medications (such as anti-hypertensive medications)
  * depression that has not been on a stable medical treatment for at least 4 weeks
* Pregnancy
* Color blindness
* Allergy to chocolate, peanuts, tree nuts, egg, soy, mike, wheat
* Individuals who are or potentially may be cognitively or psychologically impaired, or who otherwise have a limited capacity to provide consent

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Working Memory (% correct) | before, 1 hour and 3 hours post beverage
  N-Back Task
Change in Response Time (milliseconds) | before, 1 hour and 3 hours post beverage
  Simple Response Time Task
Change in Short Term Memory (# correct) | before, 1 hour and 3 hours post beverage
  Hopkins Verbal Learning Task (HVLT)
Change in Mood (change in Likert scale score) | before, 1 hour and 3 hours post beverage
  Profile of Mood Status(POMS)
Change in Attention (% accuracy) | before, 1 hour and 3 hours post beverage
  Eriksen Flanker Task
Change in Executive Function (# correct) | before, 1 hour and 3 hours post beverage
  Stroop Task

SECONDARY OUTCOMES:
Change in Brain Blood Flow (ml/g/min) | 1 hour and 3 hours post beverage
  Non-invasive brain perfusion measured with arterial spin labeling magnetic resonance imaging
% Change in Heart Rate (beats/minute) | before, 1 hour and 3 hours post beverage
  pulse
% Change in Respiration (breaths/minute) | before, 1 hour and 3 hours post beverage
% Change in Blood Pressure (mmHg) | before, 1 hour and 3 hours post beverage

OTHER OUTCOMES:
% Change in Brain Connectivity (network degree) | 1 hour and 3 hours post beverage
  Measures of functional brain connectivity based on resting-state functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Laurienti, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States